CLINICAL TRIAL: NCT03936322
Title: Minimally Invasive Fetoscopic Regenerative Repair of Spina Bifida - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rodrigo Ruano (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Rodrigo Ruano, Regulatory Sponsor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-008622
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Spina Bifida; Myelomeningocele; Neural Tube Defects
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele; Neural Tube Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pregnant women diagnosed with fetal myelomeningocele (Experimental): Women subjects who are pregnant and diagnosed with myelomeningocele (MMC), also known as fetal spina bifida or neural tube defect, will undergo a minimally invasive fetoscopic repair of MMC.
  Interventions: Device: Minimally invasive fetoscopic repair of MMC

INTERVENTIONS:
Device: Minimally invasive fetoscopic repair of MMC — Uses a technique to open your belly (skin, muscles and abdomen) without opening the uterus, except for a small puncture, to repair the fetal spina bifida defect during the second trimester of pregnancy.

SUMMARY:
Researchers are studying a new minimally invasive technique (fetoscopic repair) for repair of spina bifida (MMC) during the second trimester of pregnancy. Researchers are trying to determine if this less invasive surgical approach will have less risk to the mother and at the same time adequate closure of the fetal spina bifida defect.

ELIGIBILITY:
Inclusion Criteria

* Pregnant women - maternal age 18 years or older
* Gestational age at the time of the procedure between 19 0/7 weeks and 25 6/7 weeks
* Singleton pregnancy.
* MMC diagnosis with the upper boundary located between Thoracic 1 (T1) and Sacral

  1 (S1).
* Evidence of hindbrain herniation (confirmed on MRI to have an Arnold-Chiari type II malformation).
* Absence of chromosomal abnormalities and associated anomalies.
* Normal karyotype and/or normal chromosomal microarray (CMA) by invasive testing (amniocentesis or CVS). If there is a balanced translocation with normal CMA with no other anomalies the candidate can be included.
* Family has considered and declined the option of termination of the pregnancy at less than 24 weeks.
* Family meets psychosocial criteria (sufficient social support, ability to understand requirements for this study).
* Pregnant subject capable of consenting for their own participation in this study.
* Willingness to undergo an open MMC repair, if necessary
* Parental/guardian permission (informed consent) for follow up of child after birth.

Exclusion Criteria:

* Exclusion Criteria

  * Fetal anomaly unrelated to MMC.
  * Multiple gestation
  * Declined invasive testing for karyotype (amniocentesis or CVS)
  * Severe kyphosis (defined as curvature of the spina (vertebras) higher than 30o degree measured by ultrasonography or magnetic resonance imaging).
  * Increased risk for preterm labor including short cervical length (<2.0 cm), history of incompetent cervix with or without cerclage, and previous preterm birth.
  * Placental abnormalities (previa, abruption, accreta) known at time of enrollment.
  * A body-mass index ≥40 at first prenatal visit.
  * Contraindications to surgery including previous hysterotomy (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, major myomectomy resection, or previous fetal surgery) in active uterine segment.
  * Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, uterine anomalies incompatible with fetoscopy.
  * Amniotic Fluid Index (AFI) < 6 cm if deemed to be due to fetal anomaly, poor placental perfusion or function, or membrane rupture. Low amniotic fluid volume that responds to maternal hydration is not an exclusion.
  * Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy.
  * Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patients HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment.
  * Maternal medical condition that is a contraindication to surgery or anesthesia.
  * A score of ≥ 29 on the Beck Depression Inventory (BDI) at screening
  * Maternal hypersensitivity to collagen
  * Patient does not have a support person (i.e. Spouse, partner, mother) available to support the patient for the duration of the pregnancy.
  * Inability to comply with the travel and follow-up requirements of the trial.
  * Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruano, M.D., Ph.D., Principal Investigator — University of Miami
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnant Women Diagnosed With Fetal Myelomeningocele
Started | 3
Completed | 1
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Infant Death after delivery; therefore, no further follow up occurred | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women Diagnosed With Fetal Myelomeningocele
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maternal Adverse Events
Description: Total number of maternal adverse events
Time Frame: From time of surgery until delivery (up to 21 weeks)
Measure: Number; unit: participants
Arm/Group | Pregnant Women Diagnosed With Fetal Myelomeningocele
Number analyzed (Participants) | 3
participants | 2

2. Primary Outcome: Neonatal Adverse Events
Description: Total number of neonatal adverse events
Time Frame: From the time of surgery until 28 days of life (up 25 weeks)
Measure: Number; unit: participants
Arm/Group | Pregnant Women Diagnosed With Fetal Myelomeningocele
Number analyzed (Participants) | 3
participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pregnant Women Diagnosed With Fetal Myelomeningocele
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnant Women Diagnosed With Fetal Myelomeningocele (N=3)
Placenta abruption/neonatal demise (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnant Women Diagnosed With Fetal Myelomeningocele (N=3)
premature rupture of the membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT03936322/Prot_SAP_000.pdf